CLINICAL TRIAL: NCT01921348
Title: Pilot Study to Evaluate Ear Acupressure Effects in Treating Seasonal Allergic Rhinitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Target enrollment not met within specific time period.
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Gailen D. Marshall Jr., MD PhD, Professor of Medicine and Pediatrics, Vice Chair for Research, Department of Medicine, Director, Division of Clinical Immunology and Allergy, Chief, Laboratory of Behavioral Immunology Research, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-0165
Record Dates: First submitted 2013-08-08; First posted 2013-08-13 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-05

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Hay Fever; Hayfever; Pollen Allergy; Pollinosis; Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): 34 participants will be randomized to wear acupressure pellets in the designated acupressure points and apply pressure as instructed by the study personnel.
  Interventions: Device: acupressure pellets
- Sham (Sham Comparator): 33 participants will be randomized to wear acupressure pellets in non-specific areas of the ear and apply pressure as instructed by the study personnel.
  Interventions: Device: acupressure pellets

INTERVENTIONS:
Device: acupressure pellets — The treatment group will have acupressure pellets placed in pre-determined acupressure point on the ear that relates to rhinitis.
  Other Names: Magrain Ion Pellets
  Arms: Treatment
Device: acupressure pellets — The sham group will have acupressure pellets placed in a pre-determined non-specific acupressure point on the ear that is not related to rhinitis.
  Other Names: Magrain Ion Pellets
  Arms: Sham

SUMMARY:
We hypothesize that ear acupressure will be effective in treating seasonal allergic rhinitis by changing the immune parameters and the psychological impact factors are associated with ear acupressure treatment outcome.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the clinical potential of ear acupressure in treating seasonal allergic rhinitis. We hypothesize that ear acupressure will be effective in treating seasonal allergic rhinitis by changing the immune parameters and the psychological impact factors such as expectation, stress, depression, and anxiety can moderate the ear acupressure treatment effectiveness in allergic rhinitis by influencing the immune parameters.

ELIGIBILITY:
Inclusion Criteria:

* Seasonal allergic rhinitis was diagnosed both by history and clinical examination and by the presence at positive skin prick tests
* All participants need to have at least 2 years of seasonal allergic rhinitis symptoms and a positive skin prick test to one or more pollen allergens

Exclusion Criteria:

* use of systemic corticosteroids within past 3 months period,
* active asthma,
* hearing aid usage,
* history of adhesive tape allergy,
* history of metal allergy,
* HIV,
* hepatitis B or C,
* history of hematologic, autoimmune, or malignant disease,
* pregnancy or lactation,
* ear acupressure (EAP) or acupuncture for respiratory disease within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gailen D Marshall, MD, PhD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center - Allergy, Immunology and Asthma Care Clinic, Jackson, Mississippi, United States

REFERENCES:
- [Background] Zhang CS, Yang AW, Zhang AL, Fu WB, Thien FU, Lewith G, Xue CC. Ear-acupressure for allergic rhinitis: a systematic review. Clin Otolaryngol. 2010 Feb;35(1):6-12. doi: 10.1111/j.1749-4486.2009.02067.x. PMID 20447156
- [Background] Shiue HS, Lee YS, Tsai CN, Hsueh YM, Sheu JR, Chang HH. DNA microarray analysis of the effect on inflammation in patients treated with acupuncture for allergic rhinitis. J Altern Complement Med. 2008 Jul;14(6):689-98. doi: 10.1089/acm.2007.0669. PMID 18637763
- [Background] Rao YQ, Han NY. [Therapeutic effect of acupuncture on allergic rhinitis and its effects on immunologic function]. Zhongguo Zhen Jiu. 2006 Aug;26(8):557-60. Chinese. PMID 16941973
- [Background] Petti FB, Liguori A, Ippoliti F. Study on cytokines IL-2, IL-6, IL-10 in patients of chronic allergic rhinitis treated with acupuncture. J Tradit Chin Med. 2002 Jun;22(2):104-11. PMID 12125480
- [Background] Lee MS, Pittler MH, Shin BC, Kim JI, Ernst E. Acupuncture for allergic rhinitis: a systematic review. Ann Allergy Asthma Immunol. 2009 Apr;102(4):269-79; quiz 279-81, 307. doi: 10.1016/S1081-1206(10)60330-4. PMID 19441597
- [Background] Finniss DG, Benedetti F. Mechanisms of the placebo response and their impact on clinical trials and clinical practice. Pain. 2005 Mar;114(1-2):3-6. doi: 10.1016/j.pain.2004.12.012. Epub 2005 Jan 21. No abstract available. PMID 15733625
- [Background] Benedetti F. The placebo response: science versus ethics and the vulnerability of the patient. World Psychiatry. 2012 Jun;11(2):70-2. doi: 10.1016/j.wpsyc.2012.05.003. No abstract available. PMID 22654931
- [Background] Zheng MF, Lin C, Zheng LP, He FR, Effects of acupuncture-moxibustion on monocyte Th1/Th2 cytokine in peripheral blood of patients with perennial allergic rhinitis, Journal of Acupuncture and Tuina Science 2010;8:85-88

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Sham
Started | 9 | 9
Completed | 8 | 7
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Sham | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants] — normal individuals with symptomatic allergic rhinitis whose total symptom scores were assessed before and after the intervention Population: There were no controls (i.e. non treated) individuals int his study. All participants were randomized to either an active or sham acupressure group.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 9 | 9 | 18
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (12.1) | 36.9 (12.1) | 39.4 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Rhinoconjunctivitis Quality of Life Questionnaire (Nasal Symptoms Domain Only)
Description: RQLQ is an instrument that has 28 items in 7 domains (sleep, non-rhinoconjuctivitis symptoms, practical problems, nasal symptoms, eye symptoms activity limitations and emotional function). Participants are asked to recall impairments experienced during the previous week and to respond to each item on a 7-point scale (0=no impairment; 6=maximum impairment).
  In this protocol, we used the nasal symptoms domain only; 4 questions, total scale ranges from 0 minimum to 24 maximum.
  Longitudinal changes of nasal symptoms domain total were reported from baseline to 8 weeks.
Time Frame: 8 weeks
Population: Enrollment targets were not met for both arms/groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Sham
Number analyzed (Participants) | 8 | 7
units on a scale | 2.36 (0.89) | 2.07 (1.31)

2. Secondary Outcome: Psychological Measures
Description: Effects of ear acupressure on immune biomarkers based upon psychological differences including perceived stress, anxiety, depression and worry.
Time Frame: 8 weeks
Population: Since the immune biomarker frozen blood samples were not analyzed (due to not meeting recruitment goals), the effects of ear accupressure based upon psychological differences could not be analyzed.
Arm/Group | Treatment | Sham
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Immune Biomarkers
Description: Changes in Regulatory T(Treg), Type 1 Regulatory T (Tr1), T helper 3(TH3), T helper 1(TH1), T helper 2(TH2)cells, salivary cortisol, alpha amylase, Interferon gamma(IFNg), Interleukin 4(IL4) and Interleukin 10(IL10) cytokine production from baseline to 8 weeks.
Time Frame: 8 weeks
Population: Blood samples were collected and frozen for batch analysis, but not analyzed for data since recruitment goals were not met.
Arm/Group | Treatment | Sham
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Treatment | Sham
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

LIMITATIONS AND CAVEATS:
The target number of participants needed to achieve target power and statistically reliable results was not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No